CLINICAL TRIAL: NCT04712071
Title: Effects of a Single Dose of Intravenous Ketamine on Symptoms of Gulf War Illness in 1990-1991 Gulf War Veterans
Brief Title: Ketamine in Veterans With Gulf War Illness
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Due to the COVID pandemic we could not enroll more than one subject before funding was ending.
Sponsor: Baylor College of Medicine (Other)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marijn Lijffijt, PhD, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-46289
Record Dates: First submitted 2020-11-12; First posted 2021-01-15 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Gulf War Syndrome
Keywords: Gulf War Illness; Inflammation; N-methyl-D-aspartate; ketamine
MeSH Terms: conditions — Persian Gulf Syndrome; Inflammation | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Single group, single dose, open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine (Experimental): 40 minutes intravenous infusion of 0.5 mg/kg ketamine.
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Patients with a diagnosis of Gulf War Illness using Kansas Criteria will be enrolled to receive a single 40 minute infusion of 0.5 mg/kg ketamine.
  Other Names: Ketelar

SUMMARY:
Up to one third of the 700,000 U.S. military veterans of the 1990-91 Gulf War have Gulf War Illness (GWI), a symptom complex characterized by a combination of chronic pain, cognitive impairment, debilitating fatigue, gastrointestinal complications, and other persistent symptoms. Epidemiologic studies of 1990-1991 Gulf War veterans have identified the short but intense combined exposure to insecticides (e.g., organophosphates, DEET, permethrin), pills with anti-nerve gas agent pyridostigmine bromide (PB), and low-level chemical nerve agents as likely candidates of GWI. Animal models have shown that these neurotoxicants could induce neuroinflammation which is marked by enhanced inflammatory cytokines, and activated microglia and astrocytes. Inflammation has been linked to GWI. Secondary effects of neuroinflammation and glia activation could be excessive glutamate-mediated neuronal activation. There is currently no treatment for symptoms of GWI. Ketamine is an N-methyl-D-aspartate receptor (NMDAR) antagonist. Besides blocking activation of NMDARs, a sub-anesthetic dose (0.5 mg/kg over 40 minutes) of ketamine could be an anti-inflammatory agent, and could protect microglia and astrocytes from being activated by inflammatory agents. This low dose of ketamine has also been shown to improve fatigue within 24 hours after a single infusion, and to improve inflammatory pain. This makes ketamine a feasible candidate for the treatment of inflammation-associated symptoms of GWI. This pilot study will examine if GWI is related to NMDAR functioning, testing effects of a single 40-minute intravenous infusion of 0.5 mg/kg of ketamine on GWI symptom severity in 21 veterans of the 1990-1991 Gulf War who meet Kansas case definition criteria of GWI.

DETAILED DESCRIPTION:
Recruitment for this study starts after protocol approval by the BCM IRB, MEDVAMC R&D, and DoD HRPO. All study procedures are for research only.

Potential subjects will be recruited (i) from the Houston community with advertisements in local papers and social media, and with flyers at BCM and MEDVAMC; (ii) among veterans from the 1990-1991 Gulf War who participated in protocol H-40948 and who consented to be recontacted for future studies; (iii) among veterans from the 1990-1991 Gulf War who voluntarily registered in the Gulf War Registry (GWR) because of concerns of possible Gulf War Illness (GWI). Individuals under category (i) will contact us. Individuals under category (ii) will be contacted by phone or text. Individuals under category (iii) will be contacted by letter and, after a 10-day non-response, by phone. Before sending a letter, names in the GWR will be matched with those in CPRS. If in CRPS, medical information will be reviewed to determine study eligibility; if apparently eligible, the letter will be send. If an individual is not in CPRS, the letter will be send. The letter is uploaded in section S.

For the phone call, after providing verbal consent, veterans who are interested in the study, and who did not participate in protocol H-40948, will undergo an in-depth phone pre-screen to determine eligibility. The phone pre-screen inventories symptoms of Gulf War Illness and military history with the Gulf War Military and Health Questionnaire.

This study consists of 3 phases: screening, infusion of ketamine, telephone follow-up.

For phase 1, eligible subjects will provide a urine sample for drug and pregnancy testing, undergo blood pressure testing, will undergo an EKG, will have to provide a 20 ml (2 tsp) blood sample collected for clinical labs (an additional 10 ml (2 tsp) is optional and will be banked for future research), and will visit with a study physician for a medical examination. Finally, we will go over the Gulf War Military and Health Questionnaire assessed during the phone-screen. Total time of phase 1 is 4 to 5 hours.

If qualified for the study, subjects will be scheduled for phase 2: the administration of a single intravenous infusion of 0.5 mg/kg of ketamine. For phase 2, veterans will need to fast for at least 8 hours before the infusion; they can take their medications as prescribed. At arrival at the study site, subjects have to provide a urine sample for drug and pregnancy testing. We will go over their medical information collected in phase 1 to inventory changes, and they will undergo testing of vital signs. Before the infusion at 10 am, subjects will be asked to fill out Gulf War Military and Health Questionnaire (24 hours symptoms). A baseline of possible side effects is established with the CADSS which assess dissociative states. Finally, EEG is collected from the scalp using 4-minute resting EEG (eyes-open/eyes-closed) and 15-minute passive computer paradigm with auditory 85-dB click trains. The infusion of 0.5 mg/kg ketamine is prepared by the MEDVAMC Research Pharmacy. Ketamine is dissolved in 0.9% saline in a bag of saline with a total volume of 100 mL, and administered with an infusion pump at a constant rate. An anesthesiologist will place an indwelling catheter. We will first collect an 10 ml (2 tsp) sample of blood for pro-inflammatory cytokine. Next, the catheter is used for the infusion, which lasts 40 minutes. The EEG and blood collection is repeated at 35-minutes (the peak of ketamine concentration), and again one and two hours later. Subjects will not be discharged before four hours after the end of the infusion.

For phase 3, as part of the research procedures, subjects will be contacted by telephone or telehealth services at a pre-arranged time of mutual convenience on days 1, 2 and 7 after the infusion to inventory 24-hr symptoms with the Gulf War Military and Health Questionnaire. This procedure lasts about 45 minutes to complete

ELIGIBILITY:
Inclusion Criteria:

* Military veterans who served for any period of time in the Gulf War Theater of Operations between August of 1990 and July of 1991.
* Cases must meet Kansas GWI case definition criteria.
* Understand the study as described in the informed consent form, and be able to consent for study participation.

Exclusion Criteria:

* A physical or psychiatric illness explaining GWI case definition symptoms at the discretion of the PI.
* History of seizures.
* History of ECT or deep brain stimulation.
* History of head injury with loss-of-consciousness over 15 minutes or no recollection of events.
* Unstable serious illness at the discretion of the PI or study physician, including:

  * hepatic disease
  * renal disease
  * gastroenterologic disease
  * respiratory disease,
  * cardiovascular disease (including ischemic heart disease)
  * endocrinologic disease
  * neurologic disease
  * immunologic disease
  * hematologic disease.
* Clinically significant EKG or laboratory values at the discretion of the study physician.
* Uncontrolled hypertension (systolic BP >160 mm Hg or diastolic BP >90 mm Hg).
* Family history or own history of schizophrenia or psychosis.
* For at least two weeks before ketamine infusion, use of:

  * Antibiotics
  * Antiviral medication
  * anti-inflammatory medications (including NSAIDS) for at least two weeks before ketamine infusion.
* Being pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Change in 40Hz Auditory steady state response (ASSR) EEG power | pre-treatment baseline, 35 minutes after start of infusion (close to ketamine peak) and 95 minutes after start of infusion
  The 40Hz ASSR is an electrophysiology (EEG) paradigm that presents 1-sec trains of 1-ms 85dB clicks presented at 40Hz. Outcome measure is mean power across 32 - 42Hz averaged across fronto-central electrodes that are attached in a 64-channel electrode cap that is based on a 10-10 distribution.

SECONDARY OUTCOMES:
Change in Gulf War Military and Health Questionnaire | pre-treatment baseline and days 1, 2 and 7 after the infusion
  Questionnaire developed to screen for cognitive, pain, fatigue and other Gulf War Illness symptoms. Due to its complexity, and variability, no single measure of severity addresses all possible presentations of Gulf War Illness (GWI). Therefore, we used the symptom portion of the Gulf War Military and Health Questionnaire to assess fatigue/sleep problems, somatic pain, skin abnormalities, gastrointestinal, respiratory, and neurologic/cognitive/mood symptoms, based on the Kansas GWI and CDC CMI case definitions. To assess change in current symptoms, participants are asked about the absence (0), presence, and severity (1=mild; 2=moderate; 3=severe) of the symptoms over the past 24 hours. Score range: 0-87; higher scores indicate more and/or more severe symptoms.
Change in 4 minutes resting state EEG | pre-treatment baseline, 35 minutes after start of infusion (close to ketamine peak) and 95 minutes after start of infusion
  Patients will lay quietly with eyes open for 2 minutes and eyes closed for 2 minutes to extract power of the gamma (40Hz) EEG band.Outcome measure is relative mean EEG power across 31 - 55Hz across fronto-central electrodes attached in a 64-channel electrode cap that is based on a 10-10 distribution.
Change in CADSS dissociative states scale | Pre-treatment baseline, and 1 hour, 2 hours and 4 hours after start of infusion
  The CADSS measures dissociation and psychosis-like experiences that are sometimes experienced acutely with ketamine. The CADSS has 23 clinician-administered items, each scored from 0 (not at all) to 4 (extreme). Minimal score is 0; maximum score is 92. Higher score indicate more severe dissociation and psychosis-like experiences.

OTHER OUTCOMES:
Inflammatory cytokines and metabolites of ketamine in 10 mL blood sample: Exploratory | Pre-treatment baseline, and 1 hour, 2 hours and 4 hours after start of infusion
  This sample will be used for future study to examine acute effects of ketamine on inflammatory cytokines and metabolites of ketamine

CONTACTS AND LOCATIONS:
Overall Officials: Marijn Lijffijt, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Marijn Lijffijt, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We have not decided yet what the best way is to share the data. The data will become available, though.